CLINICAL TRIAL: NCT04494932
Title: SLAP Repair vs. Biceps Tenodesis in Patients Under 30: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-01027
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: SLAP Tear
Keywords: SLAP Repair; Biceps Tenodesis
MeSH Terms: conditions — Shoulder Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biceps Tenodesis (Experimental)
  Interventions: Procedure: Biceps Tenodesis
- SLAP Repair (Control) (Active Comparator)
  Interventions: Procedure: Self-Locking Tenotomy

INTERVENTIONS:
Procedure: Self-Locking Tenotomy — Self-locking Tenotomy describes the surgical procedure that will be performed to treat SLAP tears.
  Other Names: SLAP Repair
  Arms: SLAP Repair (Control)
Procedure: Biceps Tenodesis — Biceps tenodesis describes the surgical procedure that will be performed to treat SLAP tears.
  Arms: Biceps Tenodesis

SUMMARY:
One of the common complaints after SLAP repair is pain and stiffness. However, the more recently-described Biceps Tenodesis for SLAP tears improves upon this by addressing the long head of biceps which is thought to be the pain sources. However, only one small prior RCT has evaluated this, finding minimal difference. Both procedures are currently considered standard of care, and are decided upon based on patient and surgeon preference.

This will be a single-center randomized controlled trial. The study is comparing SLAP repair and biceps tenodesis in patients under 30 undergoing surgery for SLAP tears. The purpose of the proposed study is to evaluate the effect of SLAP repair versus biceps tenodesis in the management of SLAP tears in patients under 30 years old.

DETAILED DESCRIPTION:
Superior-labrum anterior to posterior (SLAP) tears were first described by Andrews et al. in 1985, and have been reported to be present in up to 26% of shoulder arthroscopies. While the exact cause of SLAP tears is unknown, they are often related to traumatic events and sports activity, particularly overhead sports such as baseball. Type II SLAP tears, which are characterized by superior labral fraying with a detached biceps anchor, are the most common subtype, based on the classification by Snyder et al. Treatment options include SLAP repair, biceps tenodesis, biceps tenotomy, and debridement.

One of the common complaints after SLAP repair is pain and stiffness. However, the more recently-described Biceps Tenodesis for SLAP tears improves upon this by addressing the long head of biceps which is thought to be the pain sources. However, only one small prior RCT has evaluated this, finding minimal difference. Both procedures are currently considered standard of care, and are decided upon based on patient and surgeon preference.

This will be a single-center randomized controlled trial. The study is comparing SLAP repair and biceps tenodesis in patients under 30 undergoing surgery for SLAP tears. The purpose of the proposed study is to evaluate the effect of SLAP repair versus biceps tenodesis in the management of SLAP tears in patients under 30 years old.

ELIGIBILITY:
Inclusion Criteria:

* Primary indication is for SLAP tear
* Age 18-30
* Willing and able to provide consent

Exclusion Criteria:

* Associated rotator cuff tear requiring arthroscopic repair
* Pregnant patient
* Previous shoulder surgery
* Age > 30, or < 18

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2021-12-08 (Actual)

PRIMARY OUTCOMES:
Change in Score on Visual Analogue Scale (VAS) Scale | 3 months post-op, 24 months post-op
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain possible." The total score range is 0-10. The higher the score, the higher the pain level experienced.

SECONDARY OUTCOMES:
Change in Score on American Shoulder & Elbow Surgeons (ASES) Scale | 3 months post-op, 24 months post-op
  The ASES scale consists of two subscales: pain (0-50 points) and function/disability (0-50 points), with a total score range of 0-100 points. The lower the score, the greater the pain and disability.
Change in Score on Kerlan-Jobe Orthopaedic Clinical Shoulder & Elbow (KJOC) Questionnaire | 3 months post-op, 24 months post-op
  The KJOC Score includes 10 questions with an 11-point Likert scale in the form of blocks to be ticked from 0 to 10. The total score is equal to the sum of the values of the 10 responses. The higher the score, the greater the shoulder function.
Change in Score on Shoulder Instability-Return to Sport after Injury (SIRSI) Questionnaire | 3 months post-op, 24 months post-op
  The SIRSI includes 12 questions with an 11-point Likert scale in the form of blocks to be ticked from 0 to 10. The total score is equal to the sum of the values of the 12 responses then determined in relation to 100 to obtain a percentage (0-100%). The higher the score (%), the more positive the psychological response.
Average timing of return to work/sport | up to 24 months post-op
Incidence of re-operations | up to 24 months post-op

CONTACTS AND LOCATIONS:
Overall Officials: Laith Jazrawi, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to use the data upon reasonable request. Requests should be directed to laith.jazrawi@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.